CLINICAL TRIAL: NCT01230775
Title: A Phase III, Randomized, Multicenter, Subject and Sponsor-blinded, Placebo Controlled Study to Compare the Efficacy and Safety of "Anagrelide Retard" Versus Placebo in "at Risk" Subjects With Essential Thrombocythaemia
Brief Title: Anagrelide Retard vs. Placebo: Efficacy and Safety in "At-risk" Patients With Essential Thrombocythaemia
Acronym: ARETA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AOP13007
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Essential Thrombocythaemia
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anagrelide retard (Experimental): Week 1:
  1x1 tablet/d of "Anagrelide retard" (1 tablet = 2mg; total dose = 2mg/d will be administered in week 1.
  Week 2 "Anagrelide retard": Dosing will be titrated up according to response (platelet reduction) to 4 mg/day (=2x1 tablet) in week 2.
  Week 3 - Week 4 "Anagrelide retard" In week 3 and 4, dose will either be increased or decreased to maintain platelets in the normal or close to normal range. The maximum dose is 4 tablets (=8mg Anagrelide) per day.
  Maintenance Phase "Anagrelide retard" During maintenance phase (month 2 - month 12) doses of treatment are adjusted at the highest tolerated level which is able to maintain the platelet count within the normal range.
  Month 2 - month 3: 2x1 tablet/d Month 3 - month 6: 3x1 tablet/d Month 6 - month 9: 4x1 tablet/d Month 9 - month 12: 4x1 tablet/d
  Interventions: Drug: Anagrelide retard
- Placebo (Placebo Comparator): Week 1:
  1. x1 tablet/d of Placebo will be administered in week 1.
     Placebo:
  2. x1 tablet/d of placebo will be administered in week 2.
  Placebo:
  In week 3 and week 4 the maximum dose is 4 tablets per day.
  Placebo:
  In order to guarantee blinding of subjects the number of placebo tablets to be taken by the subject will vary during maintenance period:
  Month 2 - month 3: 2x1 tablet/d Month 3 - month 6: 3x1 tablet/d Month 6 - month 9: 4x1 tablet/d Month 9 - month 12: 4x1 tablet/d
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anagrelide retard — Week 1:
  1x1 tablet/d of "Anagrelide retard" (1 tablet = 2mg; total dose = 2mg/d) will be administered in week 1.
  Week 2 "Anagrelide retard": Dosing will be titrated up according to response (platelet reduction) to 4 mg/day (=2x1 tablet) in week 2.
  Week 3 - Week 4 "Anagrelide retard" In week 3 and 4, dose will either be increased or decreased to maintain platelets in the normal or close to normal range. The maximum dose is 4 tablets (=8mg Anagrelide) per day.
  Maintenance Phase "Anagrelide retard" During maintenance phase (month 2 - month 12) doses of treatment are adjusted at the highest tolerated level which is able to maintain the platelet count within the normal range.
  Arms: Anagrelide retard
Drug: Placebo — Week 1:
  1. x1 tablet/d of placebo will be administered in week 1.
     Week 2
     Placebo:
  2. x1 tablet/d of placebo will be administered in week 2.
  Week 3 - Week 4
  Placebo:
  In week 3 and week 4 the maximum dose is 4 tablets per day.
  Placebo:
  In order to guarantee blinding of subjects the number of placebo tablets to be taken by the subject will vary during maintenance period:
  Month 2 - month 3: 2x1 tablet/d Month 3 - month 6: 3x1 tablet/d Month 6 - month 9: 4x1 tablet/d Month 9 - month 12: 4x1 tablet/
  Arms: Placebo

SUMMARY:
This is a multicenter, phase III, randomized, subject and sponsor-blinded, placebo-controlled study to determine the treatment effect of "Anagrelide retard" in subjects with Essential Thrombocythaemia (ET) at "defined risk" (definition of risk criteria: see Inclusion Criteria Section 5.1) The study is planned as a 2-stage procedure according to Bauer and Köhne: After recruitment of 140 subjects an interim analysis with re-assessment of sample size is planned in an adaptive manner.

As the confirmatory analysis will be based on a time-to-event evaluation (i.e. time to 1st clinically significant ET related event), there is no stipulated observation time identically applying for all subjects. Yet, with an interim analysis being performed after having recruited 140 subjects - which is expected to be reached after 1 year - the estimated observation time for a subject in stage I will also be about 1 year. (Details are explained in the section "Statistical Considerations").

Subjects will be randomized in a 1:1 ratio to one of the following two arms:

Group A: Anagrelide retard Group B: Placebo

An a priori stratification is planned for the JAK-2 mutational status. For exploratory purposes a post hoc stratification is used for obtaining covariate adjusted results, for the following other potentially predictive factors: sex, age, Factor V Leiden, and BMI.

Dosing will be started with 1 tablet per day for week 1 and will be titrated up according to response (platelet reduction) to 2 tablets in week 2. Dosing may be further increased or decreased according to platelet response in week 3 and 4. However, the maximum dose is 4 tablets (=8mg) per day. After week 4, the maximum dose to achieve optimal platelet counts (<450 G/L) should be maintained (for visit schedule see study flow chart section IV).

To verify a treatment response, platelet counts must be evaluated at every visit. The platelet count values will be withheld from the subjects for the duration of stage I or stage II respectively. The subjects have to agree explicitly to this procedure by signing the Informed Consent form.

This is a patient and sponsor-blinded clinical study. The trial medical is packaged in the blinded fashion to keep the patient unaware (blinded) towards the actual treatment group they were randomized to. The sponsor functions (including medical monitor, pharmacovigilance manager, clinical project manager, trial data manager and trial statistician) with stay blinded in the course of the study until the database lock. Randomization scheme will be prepared by an independent statistician (not otherwise involved in the study), and will be stored securely with no access to it by the sponsor functions mentioned above. The process of randomization (provision of the individual drug-allocation information to the subjects) will be carried out by a trained staff by Harrison, in adherence to the procedures to keep the other blinded functions unaware of this information (blinded). Unblinding envelopes, which contain the treatment code per patient number for identification of treatment in case when a safety-relevant unblinding needed, will be stored at the sponsor's site. At the end of the study, verification of the extent of maintaining the blind by checking if the envelopes have been broken, will take place and will be properly documented. If the sealed envelope will broken to provide treatment identification, the date of breaking the code, the initials of the person who broke the code and the reason will be stated on the envelope.

The operational details on the blinding procedures are outlined in the relevant working guidelines (ARETA Study Working Guideline for idv staff and ARETA Study Working Guideline for Harrison, each in its current version).

Investigator will not be blinded in this study, i.e. in case of a medical need individual patient management will be driven by the full knowledge of the trial related interventions. For the case, the sponsor will need to unblind a patient (e.g. due to safety reasons), the above mentioned (in this section) envelopes will be used.

Only treatment naïve subjects, in respect to cytoreductive drugs with confirmed diagnosis of ET (centralized re-evaluation according to WHO, 2008; see Section 6.2.1) and assessment of JAK-2 status (centralized re-evaluation of JAK-2 status; see Section 6.2.2) will be enrolled.

As described above, stage I of the study will be considered as closed as soon as 140 subjects have been recruited. The duration of stage II depends on the result of the re-assessment of sample size.

Once stage I is finished, stage I subjects will enter into an extension period for a maximum of three years.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent prior to any study specific procedures and able to comply with this protocol
2. Male or female subjects aged between 18 and 60 years,
3. Confirmed diagnosis of ET according to WHO-criteria 2008 (Appendix A) including assessment of JAK-2 status (central re-evaluation).
4. Presence of predisposing risk factors for ET related events confirmed by clinical or laboratory results:

Definition of subjects with potential risk for ET-related Events:

- Platelet count < 1.000 G/L

Additionally at least ONE of the following criteria has to be fulfilled:

* Subjects aged between 40 and 60 years or
* Subjects with ET and disease duration > 3 years (Diagnosis of ET has to be at least 3 years ago and confirmed at time of screening) or
* Subjects with ONE of the following risk factors for thrombotic complications:

  * JAK- 2 positivity
  * Protein C and/or Protein S deficiency
  * Antithrombin III deficiency
  * Factor V Leiden or Prothrombin mutation
  * Cardiovascular risk factors:
* Essential hypertension,
* Smoking (>5 cigarettes/d),
* Obesity (BMI>30),
* Cholesterol (HDL/LDL ratio < 4),
* Hormone replacement therapy,
* Hormonal contraception.

Exclusion Criteria:

1. Diagnosis of any other myeloproliferative disorder
2. High-risk status (age > 60 years, platelet count ≥ 1.000 G/L, increase of platelet count > 300 G/L within 3 month, history of thrombotic/haemorrhagic or ischemic complications).
3. Any known cause for a secondary thrombocytosis
4. Previous or current treatment of ET with cytoreductive therapy
5. Diagnosis of any malignancy, apart from ET, within the last 3 years
6. Known or suspected intolerance to the investigational product
7. Known or suspected congestive heart failure
8. WBC ≥ 15 G/L
9. Severe renal impairment (creatinine clearance <30 ml/min)
10. Severe liver impairment (ALT or AST >5 times normal)
11. Clinically significant abnormal laboratory values (excluding markers of essential thrombocythaemia)
12. Poorly controlled diabetes mellitus
13. Infection with hepatitis B, hepatitis C or HIV
14. Subjects with a history of drug/alcohol abuse (within the previous 2 years)
15. Participation in another investigational study within 6 months prior to enrolment or for a longer duration if specified in local regulations
16. Women of childbearing potential with inadequate contraception
17. Pregnant or lactating women (pregnancy test to be assessed within 7 days prior to study treatment start)
18. Any significant psychiatric disorder that, in the opinion of the investigator, might prohibit the understanding and giving of informed consent or that might prevent the subject from completing the trial.

Women of childbearing potential with inadequate contraception; women with child-bearing potential, receiving oral hormone contraception and aiming to participate in the study, will have to apply an additional effective method of contraception during the study period; male subjects, receiving investigational medicinal product, which have sexual intercourse with females of childbearing potential, should use medically acceptable and reliable method of contraception to prevent pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2010-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time to 1st clinically significant ET related event | beginning 2012

SECONDARY OUTCOMES:
Efficacy and safety | end 2013
  Efficacy
  * reduction of platelet counts
  * occurrence of change to "high risk" status (i.e. platelets > 1.000 G/L or occurrence of an ET related event)
  * number of subjects achieving a complete response
  Safety
  * Adverse Events
  * cardiovascular safety (assessed by ECG, ECHO, NT-proBNP or BNP)
  Quality of Life: SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grohmann-Izay, MD, Study Director — AOP Orphan Pharmaceuticals AG
Locations (37):
- Austria (5):
  - Uniklinik Innsbruck, Innsbruck
  - Universitätsklinik für Innere Medizin III, Universitätsklinikum Salzburg, Salzburg
  - Hanusch Krankenhaus, Vienna
  - Sozialmedizinisches Zentrum Ost, Vienna
  - Uniklinik für Innere Medizin I, Vienna
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment "Dr Georgi Stranski", Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv
  - Multiprofile Hospital for Active Treatment, "Tokuda Hospital Sofia", Sofia
  - National Specialized Hospital for Active Treatment of Hematological Diseases, Sofia
  - SHAT "Joan Pavel", Sofia
- Clinical Hospital Dubrava, Zagreb, Croatia
- Lithuania (2):
  - Kauno Medicinos Universiteto Klinikos, Kaunas
  - Klaipeda Hospital, Klaipėda
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SP Szpital Kliniczny im. A. Mieleckiego, Katowice
  - Wojewódzki Szpital Specjalistyczny, Rzeszów
  - Specjalistyczny Szpital Miejski, Torùn
  - Klinika Hematologiczna, Instytut Hematologii i Transfuzjologii, Warsaw
  - Samodzielny Publiczny Centralny Szpital, Warsaw
- Romania (6):
  - Clinical County Hospital "Dr. Constantin Opris", Baia Mare
  - "Coltea" Clinic Hospital, Bucharest
  - "Fundeni" Clinical Institute, Bucharest
  - University Emergency Hospital, Bucharest
  - Emergency County Clinic Hospital, Sibiu
  - Emergency County Hospital Târgu Mureș, Târgu Mureş
- Russia (6):
  - State Medical Institution Territorial Clinical, Krasnodar
  - Haematology Research Center of RAMS, Moscow
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Russian scientific Research Institute for Hematology and Transfusiology, Saint Petersburg
  - Saint Petersburg State Institution of Healthcare, Saint Petersburg
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
- University Hospital Bratislava, Bratislava, Slovakia
- Ukraine (5):
  - Institute of Urgent and Recovery Surgery n.a., Donetsk
  - Kmelnitskiy Regional Hospital, Khmelnitskiy
  - Institute of Haematology and Transfusiology, Kiev
  - Scientific Center of Radiation Medicine AMS of Ukraine, Kiev
  - Lviv Blood Pathology Institute, Lviv